CLINICAL TRIAL: NCT01690624
Title: A Phase I, Open-label, Cohort Dose Escalation Trial With BI 836858 in Patients With Refractory or Relapsed Acute Myeloid Leukemia and Patients With Acute Myeloid Leukemia in Complete Remission With High Risk to Relapse.
Brief Title: BI 836858 Dose Escalation in Patients With Refractory or Relapsed Acute Myeloid Leukemia and in Patients With AML in Complete Remission With High Risk to Relapse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1315.1
Record Dates: First submitted 2012-09-13; First posted 2012-09-24 (Estimated); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2024-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — BI 836858

ARMS (4):
- BI836858 10milligram(mg)(Patients with relapsed\refractoryAML) (Experimental): Patients with relapsed\refractory AML were administered BI 836858 10 mg solution for infusion intravenously on day 1 and day 8 of the 14-day cycles (1 cycle with 2 administrations).
  Interventions: Drug: BI 836858
- BI 836858 20 mg (Patients with relapsed\refractory AML) (Experimental): Patients with relapsed\refractory AML were administered BI 836858 20 mg solution for infusion intravenously on day 1 and day 8 of the 14-day cycles (1 cycle with 2 administrations).
  Interventions: Drug: BI 836858
- BI 836858 40 mg (Patients with relapsed\refractory AML) (Experimental): Patients with relapsed\refractory AML were administered BI 836858 40 mg solution for infusion intravenously on day 1 and day 8 of the 14-day cycles (1 cycle with 2 administrations).
  Interventions: Drug: BI 836858
- BI 836858 40 mg (Patients with AML in CR) (Experimental): Patients with AML in complete remission (CR) with high risk to relapse were administered BI 836858 40 mg solution for infusion intravenously on Day 1 of Cycles 1, 2 and 3. From the 4th administration onwards, patients received monthly (every second cycle) infusions (i.e. 4th infusion on Cycle 5 Day 1, 5th infusion on Cycle 7 Day 1, etc.) for overall up to 12 months of treatment unless the patient relapsed or infusions were not tolerated.
  Interventions: Drug: BI 836858

INTERVENTIONS:
Drug: BI 836858 — Monotherapy with BI 836858 administered as intravenous infusion

SUMMARY:
Patients with acute myeloid leukemia who experience a relapse after at least one prior regimen may be enrolled in this trial. In addition, acute myeloid leukemia patients who are in complete remission with high risk to relapse may be eligible for this trial. The trial will examine whether monotherapy with BI 836858 is safe and tolerable at escalating dose levels.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of relapsed or refractory AML with at least one prior treatment for acute myeloid leukemia and patients with diagnosis of acute myeloid leukemia in complete remission with high risk to relapse.
2. Expression of CD33 on more than 30% of bone marrow blasts at screening for patients with refractory or relapsed acute myeloid leukemia is required. CD33 positive expression of bone marrow blasts at the time of initial acute myeloid leukemia diagnosis is sufficient for those patients in complete remission with high risk to relapse.
3. Eastern Cooperative Oncology Group Performance Status 0, 1 or 2
4. Age 18 years or older
5. Written informed consent which is consistent with International Conference on Harmonization, Good Clinical Practice (ICH-GCP) guidelines and local legislation.

Exclusion criteria:

1. Patients with acute promyelocytic leukemia according to WHO definition.
2. Patients with refractory or relapsed acute myeloid leukemia > 5.000 blasts in the peripheral blood.
3. Anti-leukemia therapy within two weeks before first treatment with BI 836858, 4 weeks for biologics. Parallel treatment with Hydroxyurea ia allowed with refractory or relapsed acute myeloid leukemia patients.
4. Allogeneic stem cell transplantation within the last 28 days before first treatment with graft versus host disease requiring more than 20 mg of steroids per day. Steroid dosage must be stable within two weeks prior to start of treatment.
5. Patients who are candidates for allogeneic stem cell transplantation (for patients with refractory or relapsed acute myeloid leukemia).
6. Second malignancy currently requiring active therapy.
7. Symptomatic central nervous system involvement
8. Aspartate amino transferase (AST) or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (ULN), or AST or ALT greater than 5 times the ULN for those with Gilbert syndrome.
9. Prothrombin time (PT) >1.5 x ULN for subjects not on therapeutic vitamin K antagonists (phenprocoumon, warfarin)
10. Bilirubin greater than 1.5 mg/dl (>26 µmol/L) unless elevation is thought to be due to hepatic infiltration by AML, Gilbert syndrome, or hemolysis.
11. Serum creatinine greater than 2.0 mg/dl
12. Known human immunodeficiency virus (HIV) infection or active hepatitis B virus or hepatitis C virus infection.
13. Concomitant intercurrent illness, or any condition which in the opinion of the Investigator, would compromise safe participation in the study, e.g. active severe infection, unstable angina pectoris, new onset of exacerbation of a cardiac arrhythmia
14. Psychiatric illness or social situation that would limit compliance with trial requirements
15. Concomitant therapy, which is considered relevant for the evaluation of the efficacy or safety of the trial drug
16. Female patients of childbearing potential who are sexually active and unwilling to use a medically acceptable method of contraception during the trial and for 6 months after the last administration of BI 836858
17. Male patients with partners of childbearing potential who are unwilling to use condoms in combination with a second effective method of contraception during the trial and for 6 months after the last administration of BI 836858
18. Pregnant or nursing female patients
19. Treatment with another investigational agent under the following conditions:

    1. Within two weeks (4 weeks for biologics or 5 half-lives, whichever is longer) of first administration of BI 836858; or
    2. Patient has persistent toxicities from prior anti-leukemic therapies which are determined to be relevant by the Investigator.
    3. Concomitant treatment with another investigational agent while participating in this trial.
20. Prior treatment with a CD33 antibody
21. Patient unable or unwilling to comply with the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-09-13 (Actual); Primary Completion 2018-05-21 (Actual); Study Completion 2018-05-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (5):
- United States (5):
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to:
  https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Phase1, open-label, non-randomized, dose-escalation, 3+3 design study followed by expansion cohort with two separate patient populations:1) patients diagnosed with relapsed or refractory acute myeloid leukemia (AML) who have failed at least one prior line of therapy(2) patients with AML who are in complete remission (CR) with high risk to relapse.
Pre-assignment Details: This study initially enrolled patients diagnosed with refractory or relapsed AML who had failed at least 1 prior line of therapy and was later amended to include patients with AML who were in CR with a high risk to relapse.
Period: Overall Study
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Started | 12 | 8 | 7 | 3
Completed | 0 | 0 | 0 | 0
Not Completed | 12 | 8 | 7 | 3
Not completed — PD based on IWG criteria or clinical PD | 8 | 5 | 2 | 0
Not completed — Adverse event (other than DLT) | 3 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0
Not completed — Sponsor is ending trial | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 1 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Treated Set (TS): TS included patients treated with at least 1 dose of BI 836858.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR) | Total
Number analyzed (Participants) | 12 | 8 | 7 | 3 | 30
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.0 (12.4) | 60.8 (7.6) | 72.3 (6.7) | 49.0 (17.5) | 62.4 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 4 | 1 | 13
  Male | 6 | 6 | 3 | 2 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 5 | 7 | 3 | 16
  Unknown or Not Reported | 11 | 3 | 0 | 0 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 2 | 0 | 0 | 2
  White | 12 | 6 | 6 | 3 | 27
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Determination of the Maximum Tolerated Dose (MTD) of BI 836858
Description: This trial was discontinued prior to reaching the primary endpoint of determining MTD.
Time Frame: From the first administration of BI 836858 to start of the fifth administration, excluding the day of fifth administration, up to 28 days.
Population: MTD evaluable set (non-replaced patients) defined as patients who completed the first two treatment cycles.
Measure: Number; unit: Milligram (mg)
Groups:
- BI 836858 (Patients With Relapsed\Refractory AML): Comprises all dose cohorts during the dose escalation phase. Patients with relapsed\refractory AML were administered BI 836858 40 mg solution for infusion intravenously on day 1 and day 8 of the 14-day cycles (1 cycle with 2 administrations).
Arm/Group | BI 836858 (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 27 | 3
Milligram (mg) | NA — No dose limiting toxicity (DLT) events were observed in the highest dose levels studied, therefore, MTD could not be determined | NA — No DLT events were observed in the highest dose levels studied, therefore, MTD could not be determined

2. Primary Outcome: Number of Patients With Dose Limiting Toxicity (DLT) During MTD Evaluation
Description: Dose limiting toxicity was defined as any non-disease-related, non-hematological Adverse Events (AE) of Common Terminology Criteria for AE (CTCAE) grade 3 or higher. Number of patients with DLT during the MTD evaluation period for evaluation for patients with refractory or relapsed acute myeloid leukemia, the first 2 cycles (i.e. patient received at least 4 administrations of BI 836858 and reached end of Cycle 2) and for AML patients in CR with high risk to relapse, the first 2 cycles (i.e. patient has received at least 2 administrations of BI 836858 and reached end of Cycle 2).
Time Frame: as for outcome 1
Population: MTD evaluable set (non-replaced patients) defined as patients who completed the first two treatment cycles.
Measure: Count of Participants; unit: Participants
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 12 | 8 | 7 | 3
Participants | 2 | 0 | 0 | 0

3. Secondary Outcome: Best Overall Response According to International Working Group (IWG) Criteria Categorized as CompleteRemission(CR), CR With Incomplete Blood Recovery (CRi), PartialRemission (PR), TreatmentFailure (TF) and ProgressiveDisease (PD)
Description: BOR for patients with refractory/relapsed acute myeloid leukemia defined as: -CR:Morphologically leukemia free state/absolute neutrophil count≥1000/microliter(μL)and platelets≥100,000/μL. No transfusion for 1week prior to assessment -CRi:Met criteria for CR, except absolute neutrophils<1000/μl/platelets<100,000/μl -PR:Met criteria for CR, except leukemic blasts in bone marrow may range from 5 to 25% as long as count has decreased by at least 50% from pre-study treatment, or<5% blasts in presence of Auer rods or abnormal morphology -TF:Patient survives≥7 days following completion of initial 2 treatment cycles with persistent leukemia in the last peripheral blood smear or bone marrow or with persistent extramedullary disease - PD:Patient survives>7 days following completion of initial 2 treatment cycles with increase of blast population in bone marrow or peripheral blood by>50% or aggravation or new development of extramedullary disease or further deterioration or death due to leukemia
Time Frame: From first administration of study drug until the earliest of progressive disease (PD), death or last adequate disease assessment before new anti-cancer therapy, up to 299 days.
Population: Treated Set (TS): TS included patients treated with at least 1 dose of BI 836858. Only patients with relapsed/refractory AML were planned to be analysed for this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML)
Number analyzed (Participants) | 12 | 8 | 7
Participants
  CR | 0 | 0 | 0
  CRi | 0 | 0 | 0
  PR | 0 | 0 | 0
  TF | 3 | 2 | 2
  PD | 8 | 5 | 3
  Not evaluable | 1 | 0 | 1
  No assessment post-baseline | 0 | 1 | 1

4. Secondary Outcome: Progression Free Survival for Patients With Refractory or Relapsed Acute Myeloid Leukemia
Description: Progression-free survival was defined as the time from first treatment with BI 836858 until disease progression, relapse or death.
Time Frame: From first administration of study drug until progressed according to disease assessment, relapse, or death without progression, up to 167 days.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML)
Number analyzed (Participants) | 12 | 8 | 7
Days | 27.5 [17.0 to 64.0] | 29.5 [8.0 to 59.0] | 50.0 [25.0 to NA] — NA = This was not estimable due to insufficient number of patients with event

5. Secondary Outcome: Time to Treatment Failure for Patients With Refractory or Relapsed Acute Myeloid Leukemia
Description: Time to treatment was defined as the time from first treatment with BI 836858 until disease progression, relapse or death or start of next AML therapy.
Time Frame: From first administration of study drug until progressive disease, relapse, death or start of next anti-AML therapy, up to 167 days.
Population: as for outcome 3
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML)
Number analyzed (Participants) | 12 | 8 | 7
Days | 27.5 [17.0 to 32.0] | 29.5 [8.0 to 59.0] | 40.5 [25.0 to 64.0]

6. Secondary Outcome: Progression Free Survival for AML Patients in CR With High Risk to Relapse
Description: Progression-free survival was defined as the time from first treatment with BI 836858 until disease progression, relapse or death for AML patients in CR with high risk to relapse.
Time Frame: From first treatment with study drug until disease progression, relapse or death for AML patients in CR with high risk to relapse, up to 409 days.
Population: Treated Set (TS): TS included patients treated with at least 1 dose of BI 836858. Only AML patients in CR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 3
Days | NA [NA to NA] — NA = This was not estimable due to insufficient number of events

7. Secondary Outcome: Time to Treatment Failure for AML Patients in CR With High Risk to Relapse
Description: as for outcome 5
Time Frame: From first treatment with study drug until disease progression, relapse, death or start of next AML therapy for AML patients in CR with high risk to relapse, up to 409 days.
Population: TS. Only patients in CR were included in the analysis.
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 3
Days | NA [NA to NA] — NA = This was not estimable due to insufficient number of events

8. Secondary Outcome: Maximum Measured Plasma Concentration (Cmax)
Description: Maximum measured plasma concentration (Cmax) after the first infusion is presented.
Time Frame: At 5 minutes (min) before start of BI 836858 infusion and at 5 hours (hrs), 6 hrs, 9 hrs, 24 hrs and 72 hrs after BI 836858 infusion.
Population: PK parameter analysis set (PKS): This patient set includes all patients in the treated set (TS) who provide at least one pharmacokinetics (PK) parameter.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per millilitre (ng/ml)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 12 | 6 | 7 | 3
nanograms per millilitre (ng/ml) | 873 (207) | 3270 (35.4) | 6100 (82.1) | 9640 (55.7)

9. Secondary Outcome: Time From Dosing to the Maximum Plasma Concentration (Tmax)
Description: Time from dosing to the maximum plasma concentration (tmax) after the first infusion is presented.
Time Frame: as for outcome 8
Population: as for outcome 8
Measure: Median (Full Range); unit: hours (hrs)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 12 | 6 | 7 | 3
hours (hrs) | 4.43 [3.00 to 7.00] | 6.07 [5.00 to 8.80] | 5.87 [5.00 to 8.45] | 5.92 [5.18 to 6.17]

10. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval of One Week (AUC0-168)
Description: Area under the plasma concentration-time curve over the time interval of one week (AUC0-168) after the first infusion is presented.
Time Frame: At 5 minutes (min) before start of BI 836858 infusion and at 5 hours (hrs), 6 hrs, 9 hrs, 24 hrs, 72 hrs and 168 hrs after BI 836858 infusion.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/millilitre (ng*h/ml)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 12 | 6 | 7 | 3
nanograms*hours/millilitre (ng*h/ml) | NA (NA) — NA=Values below level of detection | NA (NA) — NA=Values below level of detection | NA (NA) — NA=Values below level of detection | 783000 (37.3)

11. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval of One Treatment Cycle (AUC0-tz)
Description: Area under the plasma concentration-time curve over the time interval of one treatment cycle (AUC0-tz) is presented.
  One treatment cycle included a first and a second infusion.
Time Frame: At approximately 5 minutes (min) before start of first (Day 1) and second (Day 8) BI 836858 infusion and at 5 hours (hrs), 6 hrs, 9 hrs, 24 hrs, 72 hrs and 168 hrs after first and second BI 836858 infusion.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/millilitre (ng*h/ml)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 12 | 8 | 7 | 3
nanograms*hours/millilitre (ng*h/ml)
  first infusion: number analyzed (Participants) | 12 | 6 | 7 | 3
  first infusion | 7730 (631) | 68100 (89.4) | 190000 (194) | 807000 (38.1)
  second infusion: number analyzed (Participants) | 9 | 7 | 6 | 0
  second infusion | 7980 (417) | 28100 (133) | 361000 (32.8) |

12. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero Extrapolated to Infinity (AUC0-infinity)
Description: Area under the plasma concentration-time curve over the time interval from zero extrapolated to infinity (AUC0-infinity) is presented.
Time Frame: At 5 minutes (min) before start of the first BI 836858 infusion at Day 1 and at 5 hours (hrs), 6 hrs, 9 hrs, 24 hrs and 72 hrs after the first BI 836858 infusion.
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/millilitre (ng*h/ml)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 7 | 5 | 7 | 3
nanograms*hours/millilitre (ng*h/ml) | 23400 (137) | 97900 (114) | 296000 (256) | 1120000 (39.8)

13. Secondary Outcome: Terminal Half-life (t1/2)
Description: Terminal half-life (t1/2) is presented.
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hrs)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 7 | 5 | 7 | 3
hours (hrs) | 11.3 (64.3) | 21.4 (91.7) | 34.5 (107) | 94.3 (22.1)

14. Secondary Outcome: Mean Residence Time After Intravenous Infusion (MRT)
Description: Mean residence time after intravenous infusion (MRT) is presented.
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours (hrs)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 7 | 5 | 7 | 3
hours (hrs) | 16.4 (62.1) | 30.8 (85.4) | 50.8 (98.7) | 136 (22.3)

15. Secondary Outcome: Total Plasma Clearance (CL)
Description: Total plasma clearance (CL) is presented.
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: millilitre/minute (ml/min)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 7 | 5 | 7 | 3
millilitre/minute (ml/min) | 7.11 (137) | 3.40 (114) | 2.25 (256) | 0.595 (39.8)

16. Secondary Outcome: Apparent Volume of Distribution During the Terminal Phase (Vz)
Description: Apparent volume of distribution during the terminal phase (Vz) is presented.
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (l)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 7 | 5 | 7 | 3
Litre (l) | 6.99 (51.9) | 6.29 (30.8) | 6.72 (63.9) | 4.85 (38.5)

17. Secondary Outcome: Volume of Distribution After Intravenous Infusion at Steady State (Vss)
Description: Volume of distribution after intravenous infusion at steady state (Vss) is presented.
Time Frame: as for outcome 12
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Litre (l)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 7 | 5 | 7 | 3
Litre (l) | 7.01 (53.0) | 6.30 (29.4) | 6.86 (69.5) | 4.85 (39.0)

18. Secondary Outcome: Area Under the Plasma Concentration-time Curve Over the Time Interval From Zero to the Time of the Last Quantifiable Data Point (AUC0-tz)
Description: Area under the plasma concentration-time curve over the time interval from zero to the time of the last quantifiable data point (AUC0-tz) is presented.
Time Frame: as for outcome 11
Population: as for outcome 8
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/millilitre (ng*h/ml)
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
Number analyzed (Participants) | 12 | 8 | 7 | 3
nanograms*hours/millilitre (ng*h/ml)
  First infusion: number analyzed (Participants) | 12 | 6 | 7 | 3
  First infusion | 7730 (631) | 68100 (89.4) | 190000 (194) | 807000 (38.1)
  Second infusion: number analyzed (Participants) | 9 | 7 | 6 | 0
  Second infusion | 7980 (417) | 28100 (133) | 361000 (32.8) |

ADVERSE EVENTS:
Time Frame: All AEs, including all-cause mortality, with an onset between start of treatment date and date of last treatment administration + the residual effect period of 30 days, date of death or date of data base lock; up to 409 days.
Description: AEs are presented for trial period.
Arm/Group | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) | BI 836858 40 mg (Patients With AML in CR)
All-Cause Mortality (participants affected / at risk) | 2/12 | 4/8 | 2/7 | 0/3
Serious Adverse Events (participants affected / at risk) | 9/12 | 8/8 | 6/7 | 1/3
Other Adverse Events (participants affected / at risk) | 12/12 | 8/8 | 7/7 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) (N=12) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) (N=8) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) (N=7) | BI 836858 40 mg (Patients With AML in CR) (N=3)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Retinal haemorrhage (Eye disorders) | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Catheter site haemorrhage (General disorders) | 1 | 0 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Death (General disorders) | 0 | 2 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 1 | 2 | 0 | 0
Abdominal abscess (Infections and infestations) | 0 | 1 | 0 | 0
Anorectal infection (Infections and infestations) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 0 | 0 | 0 | 1
Device related infection (Infections and infestations) | 0 | 1 | 0 | 0
Enterocolitis bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 3 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 1 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 0
Delirium (Psychiatric disorders) | 1 | 1 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 1 | 0 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI836858 10milligram(mg)(Patients With Relapsed\refractoryAML) (N=12) | BI 836858 20 mg (Patients With Relapsed\Refractory AML) (N=8) | BI 836858 40 mg (Patients With Relapsed\Refractory AML) (N=7) | BI 836858 40 mg (Patients With AML in CR) (N=3)
Anaemia (Blood and lymphatic system disorders) | 4 | 3 | 3 | 3
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 1 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 0 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 1 | 2 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 0 | 1
Diplopia (Eye disorders) | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 0 | 0 | 0 | 2
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 3 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Colonic fistula (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 3 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Glossodynia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 3 | 1 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 2 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0
Chills (General disorders) | 2 | 0 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1
Face pain (General disorders) | 1 | 0 | 0 | 0
Fatigue (General disorders) | 4 | 1 | 0 | 2
Malaise (General disorders) | 2 | 0 | 0 | 0
Mucosal inflammation (General disorders) | 1 | 0 | 1 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Graft versus host disease in eye (Immune system disorders) | 0 | 0 | 0 | 1
Alpha haemolytic streptococcal infection (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Device related infection (Infections and infestations) | 1 | 0 | 0 | 0
Lip infection (Infections and infestations) | 1 | 0 | 0 | 0
Lung infection (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 2 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 5 | 2 | 2 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0
Blood cholesterol increased (Investigations) | 0 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 1
Blood fibrinogen decreased (Investigations) | 0 | 0 | 0 | 1
Blood glucose increased (Investigations) | 1 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0 | 2
Neutrophil count decreased (Investigations) | 1 | 0 | 0 | 1
Platelet count decreased (Investigations) | 3 | 2 | 3 | 2
Transaminases increased (Investigations) | 0 | 0 | 1 | 0
Weight increased (Investigations) | 2 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 3 | 2 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 4 | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 0 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Hallucination (Psychiatric disorders) | 1 | 1 | 0 | 0
Illusion (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 0 | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0 | 0 | 0
Restlessness (Psychiatric disorders) | 0 | 0 | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 0 | 0 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 1
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Skin mass (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Essential hypertension (Vascular disorders) | 1 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0 | 1
Hypotension (Vascular disorders) | 1 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Discontinuation of prior anti-leukemia therapy was required at least 2 weeks before first administration of trial drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2016-04-28): https://cdn.clinicaltrials.gov/large-docs/24/NCT01690624/Prot_000.pdf
  • Statistical Analysis Plan (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT01690624/SAP_001.pdf